CLINICAL TRIAL: NCT05486468
Title: The Use of Two YUTIQ Versus Sham for Treatment of Chronic Non Infectious Intraocular Inflammation Affecting the Posterior Segment (TYNI Trial)
Brief Title: The Use of Two YUTIQ Versus Sham for Treatment of Chronic Non Infectious Intraocular Inflammation Affecting the Posterior Segment
Acronym: TYNI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Retina Associates (Other)
Collaborators: Eye Point Pharmaceuticals (Unknown); ANI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRA-TYNI-22-001
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Uveitis; Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate
MeSH Terms: conditions — Uveitis; Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate | interventions — Fluocinolone Acetonide; Drug Implants; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: 1 year, prospective, randomized, collaborative study.
Who Masked: Participant, Care Provider
Masking Description: The subject and the examining doctor will be masked to the treatment the subject receives on day 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): This group will receive two YUTIQ implants at day 1.
  Interventions: Drug: Yutiq 0.18 MG Drug Implant
- Control Arm (Sham Comparator): This group will receive two sham injections at day 1.
  Interventions: Other: Sham Injection

INTERVENTIONS:
Drug: Yutiq 0.18 MG Drug Implant — YUTIQ ® (fluocinolone acetonide intravitreal implant) 0.18 mg, for intravitreal injection
  Arms: Treatment Arm
Other: Sham Injection — Sham injection
  Arms: Control Arm

SUMMARY:
The Use of Two YUTIQ versus Sham for Treatment of Chronic Non Infectious Intraocular Inflammation Affecting the Posterior Segment (TYNI Trial)

DETAILED DESCRIPTION:
1.0 RATIONALE AND NEEDS ASSESSMENT Primary Eyepoint Drug(s): YUTIQ

Study Rationale:

The current data shows that in eyes from patients with chronic non-infectious posterior uveitis(NIPU), a single YUTIQ implant decreases the number of uveitis recurrences, led to less necessary adjunctive treatments, demonstrated less visual acuity loss, and had an acceptable side effect profile. Naturally, we asked whether two YUTIQ implants at the time of treatment would lead to an improved level of control of intraocular inflammation. We propose to evaluate the safety and efficacy of two YUTIQ implants versus two sham injections to manage inflammation associated with NIPU.

Needs Assessment:

Chronic noninfectious uveitis of the posterior segment of the eye is a visually debilitating disease to patients affected with it. Untreated or undertreated recurrent episodes of inflammation in these patients lead to permanent damage to the intraocular structures of the eye resulting in irreversible vision loss. Recent data has shown that a single YUTIQ implant demonstrated an improved level of control of intraocular inflammation, decreased frequency of uveitis flare ups, and led to less visual acuity loss compared to sham. However, there were still patients in the treatment group who had suboptimal control of their intraocular inflammation, experienced uveitis flares, and had a decrease in best-corrected visual acuity (BCVA). A study evaluating two YUTIQ implants for chronic NIPU would provide data to address whether this treatment paradigm would lead to superior outcomes and reduced treatment burden. There are currently no published prospective trials that have evaluated primary therapy with two YUTIQ implants.

In this study, we aim to compare the recurrence rate of uveitis by month 6 of two YUTIQ intravitreal implants to sha m. The clinical definition of intraocular inflammation recurrence is ( a 2 step or more increase in number of cells in the anterior chamber per high powered field (x1.6 using a 1 mm beam), ( a 2 step or more increase in vitreous haze, or ( a deterioration in BCVA of 15 letters or more. We expect a decreased rate of uveitis recurrences compared to sham. We also expect a decrease in inflammatory recurrences and increased time to first recurrence compared to prior data evaluating the use of a single YUTI Q implant.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Male or non-pregnant female in good general health at least 18 years of age, understands the language of the informed consent, and is willing and able to provide written informed consent and sign/date a health information release (HIPAA form) before any study procedures are performed.
2. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Ocular Inclusion Criteria (Study Eye):

1. Diagnosed with chronic unilateral or bilateral noninfectious posterior segment inflammation (with or without anterior uveitis) that demonstrated a clinical response to ≥1 previous corticosteroid treatment of any localized type (eg, topical steroid 2 to 4 times per day or intra- or peri-ocular injection) or systemic corticosteroid/immunosuppressant treatment with recurrence following treatment indicating chronicity according to the Investigator's judgment.
2. Presence of active posterior segment inflammation as determined by the Investigator.
3. Vitreous haze grade ≥ 2 based on the standardization of uveitis nomenclature (SUN) criteria.
4. Less than 10 anterior chamber cells/high power field determined by slit lamp examination.
5. Not planning to undergo elective ocular surgery during the study.

Exclusion Criteria:

General Exclusion Criteria:

1. Subjects with known hypersensitivity to any components of YUTIQ.
2. Female subjects who are pregnant or breastfeeding.
3. Has any acute or chronic medical disease or psychiatric condition that, in the opinion of the Investigator, would preclude participation in the study or put the subject at risk due to study treatment or procedures.

Ocular Exclusion Criteria (Study Eye):

1. History of anterior uveitis only (without associated uveitis that affected the posterior segment).
2. Presence of a vitreous hemorrhage.
3. Uveitis with infectious etiology.
4. Intraocular inflammation associated with a condition other than non-infectious uveitis (e.g., intraocular lymphoma).
5. Current infectious diseases of the cornea and conjunctiva, mycobacterial infections of the eye, or fungal diseases of ocular structures.
6. Subjects with ACIOL (Anterior Chamber Intraocular Lens) or rupture of the posterior lens capsule.
7. Diagnosis of any form of glaucoma or ocular hypertension at screening, unless the study eye is being treated with ≤2 intraocular pressure (IOP)-lowering medications and/or has been previously treated with an incisional surgical procedure resulting in stable IOP in the normal range (10 to 21 mmHg).
8. Intraocular pressure >21 mmHg or concurrent therapy at screening with >2 IOP-lowering pharmacologic agents in the study eye.
9. Any eye surgery within 12 weeks prior to Day 1 of the study.
10. Subjects who are unable to attend scheduled follow-up visits throughout the 12-month study.
11. Has a significant media opacity precluding evaluation of retina and vitreous in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of uveitis will be assessed at the 6-month visit | 6 months
  The primary endpoint of recurrence rate of uveitis will be assessed at the 6-month visit. The clinical definition of intraocular inflammation recurrence is (1) a 2-step or more increase in number of cells in the anterior chamber per high-powered field (x1.6 using a 1-mm beam), (2) a 2-step or more increase in vitreous haze, or (3) a deterioration in BCVA of 15 letters or more. In each case, the etiology of the change must be only due to noninfectious uveitis.

SECONDARY OUTCOMES:
Recurrence rate of uveitis at the 12-month visit | 12 months
  The secondary endpoints include determining the recurrence rate of uveitis at the 12-month visit, time to first uveitis recurrence, change in BCVA from baseline by ETDRS letters read at the 12-month visit, total number of necessary adjunctive treatments necessary, mean changes in CST as measured by SD-OCT, and mean changes from baseline in BCVA by ETDRS letters read. A final secondary endpoint will be to evaluate the changes in vascular leakage on FA, which will qualitatively be determined by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Retina Associates, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No